CLINICAL TRIAL: NCT06868056
Title: Pilot Randomized Controlled Trial of Food Policies to Promote Healthier Choices at Restaurants
Brief Title: Validation of Restaurant App
Acronym: VRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 855149
Record Dates: First submitted 2025-02-13; First posted 2025-03-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Disease
Keywords: chronic disease; sugar-sweetened beverages; warning labels; beverage tax
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be aware of their group assignment initially. It will be necessary to omit these details so that participants will shop for restaurant food as they would do in the real-world. We hope this minimizes the chances that the participant will purchase foods that they think the research team wants them to purchase. To conceal the study's purpose, participants will be told that we are conducting consumer market research about online shopping experiences, but will not be told that we are specifically interested in understanding the effects of food and beverage taxes, nutrition labels, and marketing restrictions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No ultra-processed food and beverage taxes, warning labels, or healthy checkout regulations (No Intervention): An online application that will mimic real-world restaurant ordering with no ultra-processed food and beverage taxes, warning labels, or healthy checkout regulations on any products
- Intervention (Suite of healthy food policies) (Experimental): An online application with a suite of healthy food policies, ultra-processed food and beverage taxes, front-of-pack nutrition labeling, and healthy check out regulations that restrict the promotion of ultra-processed products on the checkout page
  Interventions: Behavioral: Suite of healthy food policies

INTERVENTIONS:
Behavioral: Suite of healthy food policies — an online application with a suite of healthy food policies ultra-processed food and beverage taxes, front-of-pack nutrition labeling, and healthy check out regulations that restrict the promotion of ultra-processed products on the checkout page
  Arms: Intervention (Suite of healthy food policies)

SUMMARY:
Unhealthy diets significantly contribute to preventable chronic diseases among older adults. To advance the investigator's understanding of policies needed to support healthy diets, the objectives are: 1) to develop and validate an online fast food restaurant ordering application; and 2) to conduct a feasibility study for a larger randomized, controlled trial that will test healthy food policies in restaurant settings.

DETAILED DESCRIPTION:
To advance the investigator's understanding of policies needed to support healthy diets and nutrition security, the overall objectives are: 1) to develop and validate an online restaurant ordering application that will mimic a real fast-food restaurant; 2) to conduct a feasibility study for a larger randomized, controlled trial that will examine the extent to which healthy food policies like ultra-processed food and beverage taxes and warning labels as well as restrictions on checkout aisle marketing influence restaurant purchases. The development of this restaurant application will enable the investigator's to conduct rigorous experiments that can test policy changes to the online restaurant ordering environment. In the feasibility study, participants will be randomized to either: 1) control (no taxes, warning labels, or healthy checkout regulations on any products); or 2) a suite of healthy food policies (ultra-processed food and beverage taxes, front-of-pack nutrition labeling, and healthy check out regulations that restrict the promotion of ultra-processed products on the checkout page). The investigators propose recruiting 60 adults with low income who live in the Philadelphia, PA region. Participants will be recruited for a 3-week study. During week 1, they will be asked to make a purchase in person at a physical McDonald's location and text the research staff a picture of their receipt (a procedure that has have successfully used in the past). During weeks 2 and 3, they will be asked to shop once per week on the restaurant platform, which will be modeled after McDonald's online ordering site. Week 2 will be a baseline (control) week without interventions followed by Week 3, when the healthy food policy interventions will be introduced into the restaurant ordering interface. During each of the 3 weeks, participants will be given money to spend on their restaurant purchases. A restaurant delivery service (e.g., GrubHub) will be used to send participants the food they order. Participants will also complete a baseline and post-intervention survey. To begin to establish the validity of the online restaurant ordering app, investigators will examine the correlation between the total calories and sugars purchased as well as dollars spent when purchasing food in person vs. on the app. The rationale underlying the proposed research is based on the investigator's work showing that beverage taxes and warning labels greatly reduce SSB purchases. The research team's long-term goal is to understand the independent and combined effects of promising food policies to improve nutrition security and reduce nutrition-related diseases. The specific aims are:

Aim 1: To develop and validate an online restaurant ordering app that can be used to experimentally test the effects of food policies on restaurant purchases.

Aim 2: To conduct a pilot study on the feasibility of implementing healthy eating interventions and policies such as ultra-processed food and beverage taxes, warning labels, and checkout restrictions through the restaurant app.

Because the pilot study is a small-scale feasibility trial, it will generate descriptive statistics for outcomes, but they will not be formally analzyed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old.

Can adhere to the study schedule (e.g., receive a lunch on a Wednesday, Thursday, or Friday).

Household income approximately <200% of the federal poverty level (the same eligibility criterion as SNAP).

Reports consuming food from McDonald's or a similar fast-food chain at least once a month

Has regular internet access.

Has a smart phone that can take pictures.

Can travel to a McDonald's location to buy a meal with the study debit card

Exclusion Criteria:

Does not meet all of the inclusion criteria

Unable to provide consent non-English speaker

Cognitive impairment; per PIs discretion

Participant is under 18 years old

Doesn't in the greater Philadelphia area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Average total kcals purchased | Assessed weekly at completion of restaurant order over 3 weeks
  Our primary outcome at the person-week level will be the correlation between the mean number of calories purchased overall and from taxed/labeled products per person during the in-person restaurant shopping trip (Week 1) and their online restaurant order (Week 2) prior to the implementation of the healthy food policy interventions.
Average total sodium purchased | Assessed weekly at completion of restaurant order over 3 weeks
  Our primary outcome at the person-week level will be the correlation between the mean amount of sodium (mg) purchased overall and from taxed/labeled products per person during the in-person restaurant shopping trip (Week 1) and their online restaurant order (Week 2) prior to the implementation of the healthy food policy interventions
Average total added sugars purchased | Assessed weekly at completion of restaurant order over 3 weeks
  Our primary outcome at the person-week level will be the correlation between the mean amount of sodium (mg) purchased overall and from taxed/labeled products per person during the in-person restaurant shopping trip (Week 1) and their online restaurant order (Week 2) prior to the implementation of the healthy food policy interventions
Average total saturated fat purchased | Assessed weekly at completion of restaurant order over 3 weeks
  Our primary outcome at the person-week level will be the correlation between the mean amount of sodium (mg) purchased overall and from taxed/labeled products per person during the in-person restaurant shopping trip (Week 1) and their online restaurant order (Week 2) prior to the implementation of the healthy food policy interventions

SECONDARY OUTCOMES:
Assessing acceptability and realism of online restaurant app | Assessed at study completion, average of 3 weeks.
  We will also assess the acceptability of the online restaurant (e.g., overall experience using the restaurant, ease of use) and realism of the restaurant (e.g., extent to which participants' selections are similar to usual purchases, extent to which it felt real).
Average total dollars spent | Assessed weekly at completion of restaurant order over 3 weeks
  Our primary outcome at the person-week level will be the correlation between the mean amount of dollars spent overall and from taxed/labeled products per person during the in-person restaurant shopping trip (Week 1) and their online restaurant order (Week 2) prior to the implementation of the healthy food policy interventions

CONTACTS AND LOCATIONS:
Overall Officials: Christina Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No